CLINICAL TRIAL: NCT02238470
Title: Intracerebral Hemorrhage Due to Oral Anticoagulants in the Secondary Prevention of Ischemic Stroke: Prediction of the Risk by the Detection of Leukoaraiosis and Microbleeding With Magnetic Resonance
Brief Title: Intracerebral Hemorrhage Due to Oral Anticoagulants: Prediction of the Risk by Magnetic Resonance
Acronym: HERO
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-ACO-2010-10; PI11/00296 (Other Grant/Funding Number: FONDO DE INVESTIGACIONES SANITARIAS)
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Ischemic Stroke
Keywords: Ischemic stroke; Intracerebral hemorrhage; Subdural hemorrhage; Microbleed; Leukoaraiosis; Oral anticoagulants
MeSH Terms: conditions — Ischemic Stroke; Cerebral Hemorrhage; Hematoma, Subdural; Leukoaraiosis | interventions — Anticoagulants; Warfarin; coumarin; Dabigatran; Rivaroxaban; apixaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Oral anticoagulants: Patients who will receive oral anticoagulants indefinitely for the secondary prevention of cardioembolic stroke
  Interventions: Drug: oral anticoagulants

INTERVENTIONS:
Drug: oral anticoagulants — Comparison of patients receiving oral anticoagulants with or without microbleeds in magnetic resonance imaging
  Other Names: warfarin; coumarin; dabigatran; rivaroxaban; apixaban

SUMMARY:
The purpose of this study is to determine whether Magnetic Resonance Imaging may predict the risk of Intracerebral Hemorrhage for patients with ischemic stroke who receive indefinite oral anticoagulation

DETAILED DESCRIPTION:
OBJECTIVES. To evaluate whether Magnetic Resonance (MR) helps in predicting the risk of Intracranial Hemorrhage (ICH-OA) in patients with ischemic stroke who will receive Oral Anticoagulants (OA) for the secondary prevention of stroke. By allowing the detection and quantification of leukoaraiosis and microbleeding, MR aids in the assessment of hypertensive and/or amyloid angiopathy, two findings that may increase the risk of ICH-OA. The study of these and other known variables associated with the risk of ICH-OA will improve the selection of patients to be treated with OA. METHODOLOGY. A prospective, observational, multicentric study of 1000 patients with stroke, older than 65 y, candidates to receive OA indefinitely. The primary end-point is ICH-OA. A MR will be performed before starting the treatment, in which we will evaluate the presence and degree of leukoaraiosis (Fazekas's scale) and microbleeding (BOMBS scale). A visit will be scheduled at the first month after inclusion, and thereafter the patient will be followed-up during 2 years with phone interviews, to evaluate the appearance of the primary end-point. We will register data about demographics, vascular risk factors, anticoagulation, MR, echocardiography and co-morbidity. With those variables associated with ICH-OA in the univariate analyses, a regression analysis will be performed, in which ICH-OA will be the dependent variable. Finally, each independent predictive variable will receive a score to elaborate a predictive model of ICH-OA.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 65 y
2. TIA or ischemic stroke
3. The patient will receive indefinitely treatment with oral anticoagulants for the secondary prevention of cardioembolic stroke
4. No previous treatment with oral anticoagulants
5. Signed consent before performing a Magnetic Resonance
6. Long-term follow-up will be possible

Exclusion Criteria:

1. The patient will receive oral anticoagulation as a primary prevention treatment
2. The etiology that motivates the onset of oral anticoagulants is not cardioembolism
3. Absolute contraindication to receive oral anticoagulants
4. Arterial hypertension that is not controlled, hypertensive crisis
5. Dementia
6. Live-expectancy less than 1 year
7. Any social or psychological reason that prevents follow-up
8. Contraindication to perform a Magnetic Resonance examination
9. Patients who received oral antiacoagulants prior to the current stroke
10. The Magnetic Resonance imaging was performed more than 1 month after the onset of treatment with oral anticoagulants

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients admitted to tertiaty hospital for cardioembolic ischemic stroke
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2012-04; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Intracranial Hemorrhage | every 3 months after stroke, until 24 months
  Telephone interview every 3 months, starting 3 months after ischemic stroke (3, 6, 9, 12, 15, 18, 21 and 24 months)

SECONDARY OUTCOMES:
Ischemic stroke | within 24 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Joan Martí-Fàbregas, MD,PhD, Principal Investigator — Biomedical Research Institute Sant Pau (IIB Sant Pau)
Locations (30):
- Arcispedale Santa Maria Nuova IRCCS, Reggio Emilia, Italy
- Spain (29):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Fundació Hospital Asil Granollers, Granollers, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - Hospital Parc Taulí, Sabadell, Barcelona
  - Hospital Moisés Broggi, Sant Joan Despí, Barcelona
  - Mutua de Terrassa, Terrassa, Barcelona
  - Hospital de la Cinta, Tortosa, Tarragona
  - Hospital de Albacete, Albacete
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clínic, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital CA de Burgos, Burgos
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital de Donostia, Donostia / San Sebastian
  - Hospital Virgen de las Nieves, Granada
  - Hospital de León, León
  - Hospital Arnau de Vilanova, Lleida
  - Hospital La Rioja, Logroño
  - Hospital Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Centro Médico Asturias, Oviedo
  - Hospital Son Espases, Palma de Mallorca
  - Hospital de Navarra, Pamplona
  - CHU Santiago de Compostela, Santiago de Compostela
  - Hospital Virgen del Rocío, Seville
  - Hospital La Fe, Valencia
  - Hospital CU de Valladolid, Valladolid

REFERENCES:
- [Derived] Marti-Fabregas J, Medrano-Martorell S, Merino E, Prats-Sanchez L, Marin R, Delgado-Mederos R, Martinez-Domeno A, Camps-Renom P, Jimenez-Xarrie E, Zedde M, Gomez-Choco M, Lara L, Boix A, Calleja A, De Arce-Borda AM, Bravo Y, Fuentes B, Hernandez-Perez M, Canovas D, Llull L, Zandio B, Freijo M, Casado-Naranjo I, Sanahuja J, Cocho D, Krupinski J, Rodriguez-Campello A, Palomeras E, De Felipe A, Serrano M, Zapata-Arriaza E, Zaragoza-Brunet J, Diaz-Maroto I, Fernandez-Dominguez J, Lago A, Maestre J, Rodriguez-Yanez M, Gich I; HERO study investigators. MRI predicts intracranial hemorrhage in patients who receive long-term oral anticoagulation. Neurology. 2019 May 21;92(21):e2432-e2443. doi: 10.1212/WNL.0000000000007532. Epub 2019 Apr 19. PMID 31004066